CLINICAL TRIAL: NCT07392866
Title: A Prospective, Randomized, Active-Controlled, Open-Label, National Multicenter Phase II/III Registration Study of SH006 Injection Combination Therapy Versus Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Clinical Study of SH006 Injection in Combination Therapy Versus Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS006-II/III-01
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; immune checkpoint inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; Oxaliplatin; Capecitabine; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 SH006 in combination with bevacizumab and chemotherapy (Experimental)
  Interventions: Drug: SH006; Drug: Bevacizumab; Drug: Oxaliplatin injection; Drug: Capecitabine
- Arm 2 SH006 in combination with bevacizumab (Experimental)
  Interventions: Drug: SH006; Drug: Bevacizumab
- Arm 3 SH006 in combination with chemotherapy (Experimental)
  Interventions: Drug: SH006; Drug: Oxaliplatin injection; Drug: Capecitabine
- Arm 4 Regorafenib (Active Comparator)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: SH006 — 15 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1 SH006 in combination with bevacizumab and chemotherapy; Arm 2 SH006 in combination with bevacizumab; Arm 3 SH006 in combination with chemotherapy
Drug: Bevacizumab — 15 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1 SH006 in combination with bevacizumab and chemotherapy; Arm 2 SH006 in combination with bevacizumab
Drug: Oxaliplatin injection — 85 mg/m2 administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1 SH006 in combination with bevacizumab and chemotherapy; Arm 3 SH006 in combination with chemotherapy
Drug: Capecitabine — 1000 mg/m2 orally twice daily for 14 days continuous dosing followed by a 7-day break of each 21-day cycle
  Arms: Arm 1 SH006 in combination with bevacizumab and chemotherapy; Arm 3 SH006 in combination with chemotherapy
Drug: Regorafenib — 160 mg orally once daily for 21 days continuous dosing followed by a 7-day break of each 28-day cycle
  Arms: Arm 4 Regorafenib

SUMMARY:
To evaluate the efficacy and safety of the combination therapy of SH006 injection in the treatment of advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
This is an open, randomized, multicenter study aimed at evaluating the safety and efficacy of SH006 injection (15 mg/kg) in combination with bevacizumab and/or oxaliplatin/capecitabine versus regorafenib in the treatment of patients with advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Subjects participate voluntarily and sign informed consent.
* Age ≥ 18 and ≤ 75 years old, male or female.
* Histological or clinical diagnosis of HCC.
* Barcelona Clinic Liver Cancer stage C. BCLC stage B, not suitable for radical surgery and/or local treatment
* Previous treatment with a drug containing an immune checkpoint inhibitor failed.
* Child-Pugh ≤7 , no history of hepatic encephalopathy.

Exclusion Criteria:

* Histologically documented fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, etc.
* History of malignancy other than HCC within 5 years prior to the start of study treatment.
* History of liver transplantation, or planned to receive liver transplantation.
* Moderate or severe ascites with clinical symptoms that require drainage, uncontrolled or moderate or severe pleural and pericardical effusion.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently, or of inferior vena cava.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) (Phase II) | Up to approximately 4 years
  PFS was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Incidence of Adverse Events (AEs) (Phase II) | Up to approximately 4 years
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Overall Survival (OS) (Phase III) | Up to approximately 4 years
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 4 years
  ORR was assessed by investigators per RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR was assessed by investigators per RECIST 1.1
Duration of Response (DOR) | Up to approximately 4 years
  DOR was assessed by investigators per RECIST 1.1
Time to progression (TTP) | Up to approximately 4 years
  TTP was assessed by investigators per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Tianyinshan Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No